CLINICAL TRIAL: NCT03388307
Title: Unilateral Decompression Approach for Lumbar Canal Stenosis
Brief Title: Unilateral Approach for Bilateral Decompression of Lumbar Canal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed esam mohamed, resident doctor of neurosurgery, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29109242502338
Record Dates: First submitted 2017-12-19; First posted 2018-01-02 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unilateral laminotomy (Experimental): patients with lumbar canal stenosis who undergo unilateral laminotomy for bilateral decompression
  Interventions: Procedure: unilateral laminotomy
- decompressive laminectomy (Experimental): patients with lumbar canal stenosis who undergo decompressive laminectomy
  Interventions: Procedure: decompressive laminectomy

INTERVENTIONS:
Procedure: unilateral laminotomy — minimally invasive technique
  Arms: unilateral laminotomy
Procedure: decompressive laminectomy — classic surgery
  Arms: decompressive laminectomy

SUMMARY:
The purpose of this study was to compare standard open laminectomy with ULBD approach in regard to efficiency, safety, and clinical outcome.

DETAILED DESCRIPTION:
Lumbar stenosis is one of the common spinal pathologies; it presents with back pain, leg pain, and neurogenic claudication . Although different surgical modalities are available, the main objective of the operation is decompression of nerve roots and the spinal cord.

Minimally invasive surgical procedures and microsurgical unilateral laminotomy with bilateral spinal canal decompression (ULBD) have been reported to achieve this goal .

The objective of lumbar decompression is to decompress the neural elements while preserving stability and the spinous processes.

The object of this study is to compare outcomes following minimally invasive unilateral laminectomy for bilateral decompression (ULBD) to a standard "open" laminectomy for LSS.

ELIGIBILITY:
Inclusion Criteria:

1. age:40-80 years
2. sex:both sexes
3. symptomatic LSS with radiculopathy , neurogenic claudication , or urinary dysfunction.
4. radiologically confirmed LSS , caused by degenerative changes
5. canal stenosis at a maximum of 2 levels

Exclusion Criteria:

1. were to undergo a concomitant fusion or instrumentation placement;
2. had had previous lumbar surgeries at the same level;
3. had spondylolisthesis of any grade or degenerative scoliosis;
4. had evidence of instability on dynamic radiographs.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
back pain | one year
  visual analog scale

SECONDARY OUTCOMES:
neurogenic claudication pain | one year
  distance can be walked